CLINICAL TRIAL: NCT01324128
Title: An Open-label, Randomised, Active-controlled, Parallel Group, Multicentre, Phase 3 Study to Investigate the Safety and Efficacy of PA21 Compared With Sevelamer Carbonate Followed by a Randomised Comparison of PA21 Maintenance Dose Versus PA21-Low Dose in Dialysis Patients With Hyperphosphataemia
Brief Title: A Phase 3 Study to Investigate the Safety and Efficacy of PA21, a Phosphate Binder, in Dialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vifor Pharma (Industry)
Collaborators: Fresenius Medical Care North America (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA-CL-05A
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: PA21; Phosphate Binder
MeSH Terms: interventions — Iron; Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PA21 (2.5 g tablet) (Experimental)
  Interventions: Drug: PA21 (2.5 g tablet containing 500 mg iron)
- Sevelamer carbonate (Active Comparator)
  Interventions: Drug: Sevelamer carbonate
- PA21-1 (1.25 g tablet) (Other)
  Interventions: Drug: PA21-1 (1.25 g tablet containing 250 mg iron)

INTERVENTIONS:
Drug: PA21 (2.5 g tablet containing 500 mg iron) — Dose range of 5.0 g/day (2 tablets/day) to 15.0 g/day (6 tablets/day).
  Arms: PA21 (2.5 g tablet)
Drug: Sevelamer carbonate — Dose range of 2.4 g/day (3 tablets/day) to 14.4 g/day (18 tablets/day)
  Arms: Sevelamer carbonate
Drug: PA21-1 (1.25 g tablet containing 250 mg iron) — Low dose comparator (1.25 g/day)
  Arms: PA21-1 (1.25 g tablet)

SUMMARY:
This is a Phase 3, randomised, active controlled, multicentre study to investigate the safety and efficacy of PA21, a phosphate binder, for control of hyperphosphataemia in dialysis patients. The primary objective is to establish the efficacy of PA21 for lowering phosphate levels in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis patients with hyperphosphataemia (≥ 1.94 mmol/L; ≥ 6.0 mg/dL)
* Stable dose of phosphate binder
* Written informed consent

Exclusion Criteria:

* Hyper/hypo calcemia; hyper intact parathyroid hormone (iPTH)
* Other significant medical conditions
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1059 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Floege, MD, Principal Investigator — Medizinische Klinik II
Locations (15):
- San Antonio, Texas, United States
- LKH St. Polten, Sankt Pölten, Austria
- CHU Sart Tilman, Liège, Belgium
- Clinical Hospital Center Rijeka, Rijeka, Croatia
- Dialysis Centre Fresenius Medical Care, Sokolov, Czechia
- KfH Nierenzentrum Berlin-Neukoelln, Berlin, Germany
- Vidzemes Hospital, Valmiera, Latvia
- Vilnius University Hospital Santariskiu Clinics, Vilnius, Lithuania
- Teaching Hospital no.1 of Medical University of Lodz, Lodz, Poland
- Dialmed Clinic SRL, Sibiu, Romania
- City Mariinsky Hospital, Saint Petersburg, Russia
- Zvezdara Clinical Medical Center, Belgrade, Serbia
- Lakeview Hospital, Benoni, South Africa
- Mykolayiv Regional Hospital, Mykolayiv, Ukraine
- Dorset County Hospital NHS Foundation Trust, Dorset, United Kingdom

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Sprague SM, Ketteler M, Covic AC, Floege J, Rakov V, Walpen S, Rastogi A. Long-term efficacy and safety of sucroferric oxyhydroxide in African American dialysis patients. Hemodial Int. 2018 Oct;22(4):480-491. doi: 10.1111/hdi.12663. Epub 2018 Apr 15. PMID 29656600

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first 100HD subjects that completed Stage 1 in the PA21 treatment group entered Stage 2 and were randomised to PA21 Maintenance Dose (MD) or PA21-1 Low Dose (LD). Due to a randomisation error only 99 subjects were randomised into Stage 2.
Groups:
- PA21 Stage 1: PA21 (2.5 g tablet). Dose range of 5.0 g/day (2 tablets/day) to 15.0 g/day (6 tablets/day).
- Sevelamer Carbonate Stage 1: Sevelamer carbonate. Dose range of 2.4 g/day (3 tablets/day) to 14.4 g/day (18 tablets/day).
- PA21 (MD) Stage 2: PA21 Maintenance Dose (MD). Continuation of same dose that was being received at the end of Stage 1
- PA21-1 (LD) Stage 2: PA21-1 (1.25 g/day) Low Dose (LD) comparator for Stage 2.
Period: Stage 1
Arm/Group | PA21 Stage 1 | Sevelamer Carbonate Stage 1 | PA21 (MD) Stage 2 | PA21-1 (LD) Stage 2
Started | 710 | 349 | 0 | 0
Completed | 515 | 293 | 0 | 0
Not Completed | 195 | 56 | 0 | 0
Period: Stage 2
Arm/Group | PA21 Stage 1 | Sevelamer Carbonate Stage 1 | PA21 (MD) Stage 2 | PA21-1 (LD) Stage 2
Started | 0 | 0 | 50 | 49
Completed | 0 | 0 | 42 | 46
Not Completed | 0 | 0 | 8 | 3

BASELINE CHARACTERISTICS:
Population: For baseline characteristics, data from All Randomised patients was used.
Groups:
- Total: Total of all reporting groups
Arm/Group | PA21 Stage 1 | Sevelamer Carbonate Stage 1 | Total
Number analyzed (Participants) | 710 | 349 | 1059
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 512 | 242 | 754
  >=65 years | 198 | 107 | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (13.35) | 55.8 (14.59) | 56.2 (13.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 314 | 129 | 443
  Male | 396 | 220 | 616
Region of Enrollment [Number; unit: participants]
  United States | 345 | 171 | 516
  Europe | 159 | 77 | 236
  Russian Federation | 101 | 50 | 151
  Ukraine | 34 | 17 | 51
  Serbia | 47 | 24 | 71
  Croatia | 19 | 8 | 27
  South Africa | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Phosphorus Levels From Week 24 to Week 27
Description: Change in serum phosphorus levels compared between PA21 Maintenance Dose (MD) and PA21-1 Low Dose (LD) in Stage 2 from Week 24 to Week 27
Time Frame: Week 24, Week 27
Population: For the Primary Outcome, data from the Primary Efficacy Set (PES) was used. The PES consists of subjects who were randomized to Stage 2 and received at least 1 dose of study medication during Stage 2 and had at least 1 post-baseline (Stage 2) efficacy assessment in Stage 2.
Measure: Least Squares Mean (Standard Deviation); unit: mg/dL
Groups:
- PA21 (MD) Stage 2: PA21 Stage 2 Maintenance Dose (MD). Continuation of same dose that was being received at the end of Stage 1.
- PA21-1 (LD) Stage 2: PA21-1 Low Dose (LD) comparator (1.25 g/day) for Stage 2
Arm/Group | PA21 (MD) Stage 2 | PA21-1 (LD) Stage 2
Number analyzed (Participants) | 44 | 49
mg/dL | 0.25 (0.23) | 1.92 (0.23)

2. Secondary Outcome: Change in Serum Phosphorus Levels From Baseline to Week 12
Description: Change in serum phosphorus levels from baseline to Week 12 in the PA21 group versus the sevelamer group.
Time Frame: Week 12 post Baseline
Population: For the Secondary Outcome, data from the Per Protocol Set (PPS) was used. The PPS consists of all subjects who had completed the analysis dose titration period (baseline to Week 12), had at least 1 evaluable serum phosphorus result at or after Week 12, and had no major protocol deviations.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- PA21 (2.5 g Tablet) Stage 1: PA21 (2.5 g tablet). Dose range of 5.0 g/day (2 tablets/day) to 15.0 g/day (6 tablets/day).
Arm/Group | PA21 (2.5 g Tablet) Stage 1 | Sevelamer Carbonate Stage 1
Number analyzed (Participants) | 461 | 224
mg/dL | -2.19 (0.09) | -2.45 (0.11)

ADVERSE EVENTS:
Description: For the serious adverse event (SAE) and adverse event (AE) listings, data from the Safety Set (SS) was used. The SS consists of all randomised subjects who received at least 1 dose of study treatment.
Groups:
- PA21-1 (LD) Stage 2: PA21-1 (1.25 g tablet). Low Dose (LD) comparator (1.25 g/day) for Stage 2.
- PA21 (MD) Stage 2: PA21 (2.5g tablet) Maintenance Dose (MD). Continuation of same dose that was being received at the end of Stage 1.
Arm/Group | PA21 Stage 1 | Sevelamer Carbonate Stage 1 | PA21-1 (LD) Stage 2 | PA21 (MD) Stage 2
Serious Adverse Events (participants affected / at risk) | 129/707 | 69/348 | 6/49 | 2/45
Other Adverse Events (participants affected / at risk) | 426/707 | 162/348 | 10/49 | 2/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PA21 Stage 1 (N=707) | Sevelamer Carbonate Stage 1 (N=348) | PA21-1 (LD) Stage 2 (N=49) | PA21 (MD) Stage 2 (N=45)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 9 (9) | 0 (0) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arterial thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Arteriovenous graft (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous graft site infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ateriovenous shunt operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bactiuria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bleeding varicose vein (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood glucose abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calciphylaxis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheterisation cardiac (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 8 (9) | 5 (6) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congestive cardiac failure (Cardiac disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Diabetic eye disease (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Duodenitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Graft infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cyst infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leriche syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device complications (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 7 (7) | 2 (2) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cyst infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal transplant (Surgical and medical procedures) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 4 (5) | 3 (3) | 0 (0) | 0 (0)
Sepsis syndrome (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shunt infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shunt occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shunt stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis in device (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxic encelphalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PA21 Stage 1 (N=707) | Sevelamer Carbonate Stage 1 (N=348) | PA21-1 (LD) Stage 2 (N=49) | PA21 (MD) Stage 2 (N=45)
Diarrhoea (Gastrointestinal disorders) | 142 (184) | 26 (31) | 1 (1) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 109 (110) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 79 (114) | 27 (39) | 7 (7) | 0 (0)
Nausea (Gastrointestinal disorders) | 51 (60) | 39 (41) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 45 (54) | 26 (39) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 31 (36) | 19 (22) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 23 (25) | 7 (7) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 27 (33) | 25 (26) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators may not present or publish partial or complete study results individually. Any manuscript or abstract proposed by the Investigators must be reviewed and approved in writing by Vifor Pharma before submission for publication. Names of all Investigators participating in the study will be included in the publication.